CLINICAL TRIAL: NCT00973531
Title: Effect of Treating Sleep Disorder Breathing Therapy in Patients With Resistant Hypertension
Brief Title: Effect of Treating Sleep Disorder Breathing in Patients With Resistant Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Darshak Karia, MD, Albert Einstein Healthcare Network, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN 4113
Record Dates: First submitted 2009-09-02; First posted 2009-09-09 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Sleep Apnea; Hypertension
Keywords: Sleep Disordered Breathing; Sleep Apnea; Hypertension; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulatory APAP and SMT (Other): Subjects placed on the APAP machine
  Interventions: Device: Autotitrating Positive Airway Pressure (APAP)
- Titration Polysomnogram with CPAP and SMT (Other): Subjects placed on CPAP machine
  Interventions: Device: Traditional Split Titration Polysomnogram

INTERVENTIONS:
Device: Autotitrating Positive Airway Pressure (APAP) — Then subjects will use Autotitrating Positive Airway Pressure machine for 90 days
  Arms: Ambulatory APAP and SMT
Device: Traditional Split Titration Polysomnogram — Then subjects will use Continuous Positive Airway Pressure (CPAP) machine for 90 days
  Arms: Titration Polysomnogram with CPAP and SMT

SUMMARY:
The investigators would like to investigate the effects of treating sleep apnea with a positive airway pressure device, either continuous (titrated) versus auto titrated on the control of blood pressure in patients with Resistant Hypertension.

DETAILED DESCRIPTION:
One of the major cause and contributor to stroke, myocardial infarction, heart disease, and kidney disease is high blood pressure. Traditional approaches to control of hypertension (HTN) have mostly included pharmaceuticals targeting different mechanisms that contribute to HTN. However, adequate control of Blood pressure continues to remain a major problem.

Sleep Apnea is currently being recognized as a modifiable risk factor for resistant HTN. Sleep disordered breathing represents states of increased sympathetic drive and vagal tone withdrawal, along with significant episodic hypoxia. There is increasing evidence that sleep apnea is highly prevalent in subjects with hypertension and may be a frequent cause of drug-resistant hypertension.

We propose that we compare strategies for treating subjects with Resistant Hypertension who have SDB as detected by ambulatory multi somnogram and treat subjects using:

1. Ambulatory Autotitrating Positive Airway Pressure (APAP) plus Standard medical therapy OR
2. Traditional Polysomnogram and Traditional PSG guided titration of Continuous Positive Airway Pressure (CPAP) plus Standard medical therapy

Our hypothesis is that in subjects with Resistant HTN, who have SDB, using the treatment approach of ambulatory multisomnography for testing and then treating with APAP will be noninferior to the traditional polysomnography plus CPAP approach in the amount of reduction of mean systolic and diastolic 24 hour ambulatory blood pressure, when treated for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are competent to provide written consent
* Aged 18 to 80 years
* Deemed to be compliant with anti-hypertension medication therapy.
* Subjects with diabetes and/or chronic kidney disease must have a mean 24 hour systolic blood pressure ≥130 mmHg
* All other subjects must have a mean 24 hour systolic blood pressure ≥140 mmHg
* Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, preferably including a diuretic

Exclusion Criteria:

* Average sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg
* Known Sleep apnea
* Subjects who perform alternating shift or night work
* Subjects who have participated in a clinical study involving another investigational drug or device within 4 weeks prior to Screening
* Have hypertension secondary to an identifiable and treatable cause other than sleep apnea
* Subjects taking over the counter medications that can raise blood pressure, such as

  * Non narcotic analgesics
  * Non steroidal anti-inflammatory agents, including aspirin, Selective COX-2 inhibitors
  * Sympathomimetic agents (decongestants, diet pills, cocaine)
  * Stimulants (methylphenidate, dexmethylphenidate, dextroamphetamine, amphetamine, methamphetamine, modafinil)
  * Alcohol
  * Oral contraceptives
  * Cyclosporine
  * Erythropoietin
  * Natural licorice
  * Herbal compounds (ephedra or ma huang)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Noninferiority of the change from baseline to 90 day measurement in mean ambulatory 24-hour systolic ambulatory blood pressure in the Newer approach v/s Traditional Approach | 90 days

SECONDARY OUTCOMES:
Noninferiority of the change from baseline to 90 day measurement in mean ambulatory 24-hour diastolic ambulatory blood pressure in the Newer approach v/s Traditional Approach | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Darshak Karia, MD, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States